CLINICAL TRIAL: NCT03213171
Title: Promoting Organ and Tissue Donation Registration in Family Physician Offices: a Pragmatic Stepped-wedge Cluster Randomized Controlled Registry Trial (RegisterNow Trial)
Brief Title: Promoting Organ Donor Registration in Family Physician Offices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Institute for Clinical Evaluative Sciences (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amit Garg, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CIHR-SCT-151609
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Organ Donation; Registration for Deceased Organ Donation
Keywords: organ donation; family physician; primary care; clinical trial; registry trial; cluster trial; stepped-wedge

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care / Standard of care No intervention implemented
- Intervention (Experimental): Reception staff providing handout; Mobile tablet that provides the immediate opportunity for patients to register in the waiting room
  Interventions: Behavioral: Reception staff providing handout.; Behavioral: Mobile Tablet (e.g. iPad)

INTERVENTIONS:
Behavioral: Reception staff providing handout. — Reception staff will provide an educational pamphlet to patients that have not yet registered for organ donation
  Arms: Intervention
Behavioral: Mobile Tablet (e.g. iPad) — Patients will have the opportunity to immediately register for organ donation using an a mobile tablet (e.g. IPad)
  Arms: Intervention

SUMMARY:
This study evaluates the effects of using reception staff to prompt patients by providing a pamphlet and an opportunity to register in the waiting room via a mobile tablet on deceased organ donor registration rates.

DETAILED DESCRIPTION:
Background: There is a worldwide shortage of organs available for transplant, leading to preventable morbidity and mortality. While the majority of the general public in many countries support organ donation, actual donor registration rates are substantially out of step with these views. For instance, in Canada most Canadians support organ donation but less than 25% in most provinces have registered. The family physician office is a promising yet underused setting in which to address known barriers and facilitators to registration for deceased organ and tissue donation and to provide an immediate opportunity to register while in the waiting room for those wanting to do so.

Methods/Design: The investigators aim to evaluate the effects of having reception staff in family physician offices to prompt patients upon check-in with an educational pamphlet using a cluster, stepped-wedge randomized design. A mobile tablet will also be added to the waiting area to provide patients with the immediate opportunity to register. Family physicians are also provided with an educational booklet and encouraged to discuss organ donation with their patients. The investigators will use behaviour change techniques designed to address previously anticipated barriers and enablers to organ and tissue donation registration. The investigators will evaluate the effectiveness of the intervention conducted in six family physician offices in Ontario, Canada. Following a two-week baseline control period, offices will cross sequentially into the intervention arm in a random sequence at two-week intervals until all offices deliver the intervention (baseline + two weeks for each of six offices). The primary outcome will be the proportion of patients that have registered for deceased organ donation following in the 7 days following their office visit, using routinely collected registry data (i.e. administrative databases). The investigators will also conduct a qualitative post-trial process evaluation will assess reception staff and family physicians experiences with the intervention.

Discussion: Promoting organ and donor registration remains an important strategy for organ procurement organizations and patients worldwide. The results of this trial will inform a provincial roll-out strategy to promote organ donation in family physician offices.

ELIGIBILITY:
Inclusion/Exclusion Criteria for Patients

Inclusion Criteria:

* Patients that visited a family physician
* Patients that are at least 16 years of age with a valid health card (eligibility criteria to register for organ donation in Ontario)

Inclusion/Exclusion Criteria for Family Physicians (Cluster level)

Inclusion Criteria:

- Working at a site that sees at least 100 patients per week

Exclusion Criteria:

- Working at multiple sites that cannot be separated in analyses

Ages: 16 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Donor registration status at 7 days | 7 days
  Donor registration status (Yes/ Not registered)

SECONDARY OUTCOMES:
Donor registration status at 14 days | 14 days
  Donor registration status (Yes/ Not registered)
Donor registration status at 30 days | 30 days
  Donor registration status (Yes/ Not registered)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - City of London, London, Ontario
  - City of Stratford, Stratford, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li AH, Garg AX, Grimshaw JM, Prakash V, Dunnett AJ, Dixon SN, Taljaard M, Mitchell J, Naylor KL, Faulds C, Bevan R, Getchell L, Knoll G, Kim SJ, Sontrop J, Tong A, Bjerre LM, Hyjek K, Currie D, Edwards S, Sullivan M, Harvey-Rioux L, Presseau J. Promoting deceased organ and tissue donation registration in family physician waiting rooms (RegisterNow-1): a pragmatic stepped-wedge, cluster randomized controlled registry trial. BMC Med. 2022 Mar 3;20(1):75. doi: 10.1186/s12916-022-02266-8. PMID 35236353
- [Result] Li AH, Garg AX, Prakash V, Grimshaw JM, Taljaard M, Mitchell J, Matti D, Linklater S, Naylor KL, Dixon S, Faulds C, Bevan R, Getchell L, Knoll G, Kim SJ, Sontrop J, Bjerre LM, Tong A, Presseau J. Promoting deceased organ and tissue donation registration in family physician waiting rooms (RegisterNow-1 trial): study protocol for a pragmatic, stepped-wedge, cluster randomized controlled registry. Trials. 2017 Dec 21;18(1):610. doi: 10.1186/s13063-017-2333-5. PMID 29268758